CLINICAL TRIAL: NCT06966674
Title: Assessment of No-Reflow in Patients With STEMI After Intracoronary Tirofiban After Opening of the Track
Brief Title: No-Reflow in Patients With STEMI After Intracoronary Tirofiban After Opening of the Track
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohammed Ali Mohammed Hammad, Lecturer of Cardiology, Faculty of Medicine, Kafr Elsheikh University, Kafr Elsheikh, Egypt., Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KFSIRB200-587
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: No-Reflow; STEMI; Intracoronary; Tirofiban
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Tirofiban; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracoronary tirofiban group (Experimental): Patients will receive intracoronary tirofiban (Aggrastat®) (25 mg/kg)
  Interventions: Drug: Intracoronary tirofiban
- Control group (Placebo Comparator): Patients will receive intracoronary saline 0.9% solution as a control group.
  Interventions: Drug: Saline 0.9%

INTERVENTIONS:
Drug: Intracoronary tirofiban — Patients will receive intracoronary tirofiban (Aggrastat®) (25 mg/kg).
  Other Names: Aggrastat
  Arms: Intracoronary tirofiban group
Drug: Saline 0.9% — Patients will receive intracoronary saline 0.9% solution as a control group.
  Arms: Control group

SUMMARY:
This study aims to assess the no-reflow in patients with STEMI after intracoronary glycoprotein IIb/IIIa inhibitors after opening of track in thrombus.

DETAILED DESCRIPTION:
ST-segment-elevation myocardial infarction (STEMI) is most commonly caused by rupture or erosion of an atherosclerotic plaque, resulting in acute occlusion of the coronary artery, and the preferred reperfusion strategy is primary percutaneous coronary intervention (PCI).

The no-reflow phenomenon is one of the most common causes of adverse cardiovascular events in patients STEMI.

In recent years, mechanical or pharmacological treatment strategies including adjunctive administration of glycoprotein IIb/IIIa inhibitors (GPI) have been proposed in patients with STEMI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Both sexes.
* Patients with STEMI. ST-segment elevated myocardial infarction is defined as typical chest pain >30 minutes with ST-segment elevation of >1 mm in at least 2 consecutive leads on the electrocardiogram or new-onset left bundle brunch block.

Exclusion Criteria:

* Treatment with thrombolytic drugs in the previous 24 hours.
* Known malignancy.
* Thrombocytopenia.
* End-stage liver disease.
* Cardiogenic shock.
* Renal failure with glomerular filtration<30 ml/min.
* Contraindication for the use of tirofiban.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Blood stream | After treatment (Up to 15 minutes)
  Blood stream in coronary artery before and after treatment, including Thrombolysis in Myocardial Infarction (TIMI) flow grade in IRAs, coronary blood flow will be calculated with TIMI frame count method.

SECONDARY OUTCOMES:
Incidence of major adverse cardiac events | After treatment (Up to 30 days)
  Incidence of major adverse cardiac events were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.